CLINICAL TRIAL: NCT07216079
Title: An Open-label Extension Study for Oral Rilzabrutinib in Adults With Chronic Immune Thrombocytopenia (ITP) Who Have Completed the Long-term Extension (LTE) of the LUNA 3 Study (PRN1008 018/EFC17093) in Japan
Brief Title: Rilzabrutinib for the Adult Participants With Chronic ITP Who Have Completed Phase 3 Study in Japan
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS19407; U1111-1319-5468 (Registry Identifier: WHO)
Record Dates: First submitted 2025-10-09; First posted 2025-10-14 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rilzabrutinib (Experimental): 400 mg
  Interventions: Drug: rilzabrutinib

INTERVENTIONS:
Drug: rilzabrutinib — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: SAR444671

SUMMARY:
This is an open-label, multi-center, single group, Phase 3 study for treatment with rilzabrutinib.

The purpose of this study is to provide continuation of rilzabrutinib treatment to adult participants with ITP who have completed the LTE of the LUNA 3 study in Japan, demonstrating clinically meaningful benefit as judged by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have been enrolled in and have completed the LTE of the LUNA 3 study with demonstration of efficacy without major safety concern while on study considered by the Investigator to be clinically meaningful.
* Participants who have ongoing diagnosis of primary ITP and continue to require treatment for ITP according to the Investigator.
* Participants who have acceptable benefit/risk profile.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Participants with secondary ITP.
* Pregnant or lactating women.
* Electrocardiogram (ECG) findings for participants. The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
AEs including SAEs and AESIs | Until study completion, approximately 60 weeks
  An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor is required

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Investigational Site Number: 1001, Tsuchiura, Ibaraki
  - Investigational Site Number: 1002, Kanazawa, Ishikawa-ken
  - Investigational Site Number: 1003, Iruma-gun, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LTS19407 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26885&tenant=MT_SNY_9011